CLINICAL TRIAL: NCT06236880
Title: A Phase 2a Study to Evaluate the Safety and Tolerability of Two Repeated Doses of GM-2505 at a 2-Week Interval in Patients With Major Depressive Disorder.
Brief Title: A Phase 2a Study to Evaluate the Safety and Tolerability of GM-2505 in Patients With MDD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilgamesh Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GM-2505-201; 2023-000846-40 (EudraCT Number); M26-286 (Other: Gilgamesh Pharmaceuticals)
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Adjunctive; antidepressant; 5HT2a agonist
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose to High Dose of GM-2505 (Experimental)
  Interventions: Drug: GM-2505
- Moderate Dose to High Dose of GM-2505 (Experimental)
  Interventions: Drug: GM-2505
- Experimental very low dose to very low dose of GM-2505 (Active Comparator)
  Interventions: Drug: GM-2505

INTERVENTIONS:
Drug: GM-2505 — IV

SUMMARY:
This is a three-part Phase 2a study. The aim of Part A is to assess the safety and tolerability and preliminary antidepressant efficacy in patients with MDD who are not currently on an antidepressant therapy. The aim of Part B is to assess the antidepressant efficacy, safety and tolerability in patients with MDD who are partial responders while on a current and adequate single SSRI or SNRI treatment. Part C aims to replicate the monotherapy findings of Part A, but with a lower control group dose.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients are male or female, of any ethnic origin.
2. Patients are aged between 18 to 65 years, inclusive.
3. Patients meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for recurrent MDD without psychotic features, as assessed with the Mini-International Neuropsychiatric Interview (MINI) at Screening.
4. Current moderate to severe MDD diagnosis confirmed with a MADRS-SIGMA
5. Concomitant depression therapy:

   1. (Part A) Patients need to be stable and must not have taken any SSRI or SNRI for at least 6 weeks prior to Screening and must be willing to avoid starting a new pharmacological treatment for MDD until the end of the study procedures and assessments. Discontinuing current treatment is not allowed if done for the purposes of achieving eligibility for this study.
   2. (Part B) Patients need to be on stable treatment with any SSRI or SNRI for at least 6 weeks prior to screening and must be willing to remain on the SSRI or SNRI for the duration of the trial
   3. Patients receiving any form of psychotherapy or counselling must have been receiving therapy at Screening and must be willing to remain in therapy until the end of the study procedures and assessments.

Key Exclusion Criteria:

1. Patient has current or past primary DSM-5 diagnosis of a psychotic disorder or MDD with psychotic features, bipolar, or related disorders. A current diagnosis of PTSD, complex PTSD and borderline personality disorder are exclusionary. Other psychiatric disorders besides MDD should not be the primary disorder.
2. In first degree relatives, a history of schizophrenia, psychosis, bipolar disorder, delusional disorder, paranoid personality disorder or schizoaffective disorder.
3. Current or prior (six weeks before Screening) use of any SSRI/SNRI medication (Part A only).
4. Current or prior (five weeks before Screening) use of any monoamine oxidase inhibitor ([MAO-I]; including phenelzine, tranylcypromine, isocarboxazid, iproniazid, selegiline, rasagiline, the reversible MAO-I moclobemide and the antibiotic linezolid).or any tricyclic antidepressant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability (Part A, B, and C) | 99 Days
  The primary objective of this study is to evaluate the safety and tolerability of two doses of GM-2505 administered to MDD patients at a 2-week interval between doses.
MADRS Score (Part B and C) | 29 Days
  The estimated difference between Arm 1 and Arm 2 in the changes from baseline in MADRS-SIGMA total score

SECONDARY OUTCOMES:
MADRS-SIGMA total score (Part A) | Days 14 and 29
  Change in MADRS-SIGMA total score between Baseline and Day 29 and comparison of Day 1 low dose vs moderate dose at Day 14
MADRS-SIGMA total score (Part B and C) | All additional timepoints
  MADRS-SIGMA scores (change from baseline)
MADRS-SIGMA total score (Part B and C) | Days 14, 29, 43, 71, and 99
  Response and Remission
PK of GM-2505 (Part C) | Day 16
  Assess the pharmacokinetics of GM-2505 at very low, moderate, and high doses

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Marek, MD, Study Chair — Gilgamesh Pharmaceuticals
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom